CLINICAL TRIAL: NCT05131282
Title: An Observational Study of a Maternal Blood Protein Predictor for Case Finding of Pregnancies At Risk of Preeclampsia At Early Gestation
Brief Title: Maternal Serum Markers Predicting Preeclampsia At Early Gestations
Status: Completed | Type: Observational
Sponsor: HBI Solutions Inc. (Industry)
Collaborators: Shenzhen Maternity & Child Healthcare Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Women's Hospital, of Zhejiang University School of Medicine (Unknown); Third Affiliated Hospital of Zhengzhou University (Other); Qilu Hospital of Shandong University (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Jianmin Niu, Professor, Shenzhen Maternity & Child Healthcare Hospital
Other Study IDs: PE_001
Record Dates: First submitted 2021-10-29; First posted 2021-11-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pre-eclampsia; Preterm Birth
Keywords: pre-eclampsia; maternal serum marker; preterm pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PE group: Women with a confirmative diagnosis of PE
  Interventions: Diagnostic Test: Blood test of PE risk
- Normal pregnancy group: Normal pregnant women
  Interventions: Diagnostic Test: Blood test of PE risk; Diagnostic Test: Blood test of Preterm PE risk
- Preterm PE group: Women with a confirmative diagnosis of Preterm PE
  Interventions: Diagnostic Test: Blood test of Preterm PE risk

INTERVENTIONS:
Diagnostic Test: Blood test of PE risk — A blood test is applied to women between 11weeks and 13 weeks+6 days of GA at the first visit to evaluate risk of developing PE
  Groups: Normal pregnancy group; PE group
Diagnostic Test: Blood test of Preterm PE risk — A blood test is applied to women between 11 weeks and 13 weeks+6 days of GA at the first visit to evaluate risk of developing Preterm PE
  Groups: Normal pregnancy group; Preterm PE group

SUMMARY:
This observational study aims to assess the effectiveness of a maternal blood test as a prognostic tool for predicting early pregnancy risk of preeclampsia (PE).

We hypothesize that specific circulating protein markers may serve as reliable biomarkers for PE risk prediction. Our PE predictor is a standalone blood test designed for early gestation screening to identify pregnancies at risk. This test measures concentrations of four proteins between 11 weeks and 13 weeks+6 days of gestation.

Based on the levels of these analytes, the test generates a risk score to classify patients as either low or high risk for PE.

DETAILED DESCRIPTION:
Background and rationale:

Preeclampsia (PE) is a severe medical condition that affects 2-4% of pregnant women globally and is characterized by high blood pressure along with organ damage, particularly to the liver and kidneys. It is one of the leading causes of maternal and fetal morbidity and mortality worldwide. Early detection and preventative management of PE, including the use of low-dose aspirin, are essential for safeguarding the health of both the mother and the developing fetus. The British National Institute for Health and Care Excellence (NICE) and the American College of Obstetricians and Gynecologists (ACOG) use risk factor-based guidelines to identify women at high risk for PE. These guidelines treat each risk factor independently, leading to additive detection rates but low overall sensitivity. NICE guidelines detect only 40% of preterm PE and 35% of all PE cases with an 11% false positive rate, while ACOG detects just 5% of preterm and 2% of term PE. ACOG recommends low-dose aspirin only for women with a history of preeclampsia in multiple pregnancies or preterm delivery before 34 weeks, covering just 0.3% of all pregnancies, 5% of preterm PE, and 2% of term PE. The Fetal Medicine Foundation (FMF) PE test is utilized in several studies for screening and assessing the risk of developing PE during the first trimester. This test measures biochemical markers, such as pregnancy associated plasma protein A (PAPP-A) and placental growth factor (PlGF), in maternal blood to calculate individual risk scores. However, its limitations have highlighted the need for more effective and reliable alternatives. Performance varies across clinical sites, with sensitivity reported as low as 39-40%, and its positive predictive value (PPV) is relatively low, typically around 10-20%. This results in a significant number of false positives and negatives, which can lead to unnecessary anxiety for pregnant women and may result in missed diagnoses for those at risk. Furthermore, the FMF test requires specialized equipment and techniques, such as ultrasound for measuring the uterine artery pulsatility index (UAPI), making it less accessible in resource-limited settings and inaccuracy due to variance from different operators. These constraints limit its widespread use, underscoring the urgent need for improved blood tests to enhance prediction accuracy and reduce false results.

Clinical significance and potential impact of the test:

Advancements in medical research and technology are paving the way for more effective blood tests to improve pre-eclampsia care management. By integrating additional biomarkers and employing cutting-edge diagnostic tools such as genomics, proteomics, and metabolomics, we aim to enhance the precision and reliability of preeclampsia predictions. Our current research showcases the use of four blood serum protein markers to assess the risk of pre-eclampsia in women during early gestation (11-13 weeks), well before clinical symptoms arise.

To further validate the prediction and diagnosis performance of the novel preeclampsia test, we will enroll patients and initiate a large, multi-center observational clinical trial, including four diverse Asia cohorts, to test whether this standalone solution could bypass the need for complex maternal assessments.

Objectives and primary hypothesis of the study:

The primary objective of this study is to evaluate the predictive performance of the test for preterm preeclampsia (PE), specifically assessing its sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV). Additionally, the study aims to examine the test's predictive performance for overall PE, using the same performance metrics. We hypothesize that specific circulating protein markers may serve as reliable biomarkers for identifying pregnancies at risk for PE.

TRIAL DESIGN:

This trial is a multicenter observational study conducted in real-world clinical settings.

OUTCOMES:

The primary outcome is the diagnosis of PE during pregnancy, following the America College of Obstetricians and Gynecologists (ACOG, 2019) criteria. This diagnosis will be based on a systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg, measured on multiple occasions after 20 weeks of gestation, alongside proteinuria (dipstick urinalysis ≥ 1+ or a protein/creatinine ratio ≥ 30 mg/mmol [0.3 mg/mg]) or other signs of maternal organ dysfunction. PE will be categorized by gestational age at delivery as early-onset (<34 weeks), preterm (<37 weeks), or term (≥37 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 18 to 40 years.
2. Gestational age between 11 weeks and 13 weeks+6 days of GA at the first visit, as confirmed by ultrasound.
3. Control group: Pregnancies with no risk factors for preterm delivery, preeclampsia, or fetal growth restriction, selected during routine prenatal care between 11 weeks and 13 weeks+6 days of GA.
4. Informed consent to participate in the study.

   Exclusion Criteria:
5. Multiple pregnancies.
6. Pregestational diabetes.
7. Chronic hypertension.
8. Systemic diseases (e.g., chronic kidney disease, autoimmune disorders).
9. Any maternal or fetal condition necessitating pregnancy termination.
10. Known major fetal anomalies or fetal demise.
11. Active vaginal bleeding.
12. Serious medical illnesses (e.g., renal insufficiency, congestive heart failure, chronic respiratory insufficiency).
13. Asthma requiring systemic corticosteroids.
14. Use of anti-platelet or non-steroidal anti-inflammatory drugs.
15. Active hepatitis.
16. Lack of informed consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: A multiple-site prospective cohort of women who developed PE (i.e. the PE group) and women who had normal pregnancy (i.e. the Normal group) will be recruited. Maternal serum samples were collected between 11 weeks and 13 weeks+6 days of GA. The two group of women are matched by age, BMI, pregnant history, and other clinical information.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
diagnosis of PE during pregnancy | an average of up to 1 year
  The primary outcome is the diagnosis of PE during pregnancy, following the America College of Obstetricians and Gynecologists (ACOG, 2019) criteria. This diagnosis will be based on a systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg, measured on multiple occasions after 20 weeks of gestation, alongside proteinuria (dipstick urinalysis ≥ 1+ or a protein/creatinine ratio ≥ 30 mg/mmol [0.3 mg/mg]) or other signs of maternal organ dysfunction. PE will be categorized by gestational age at delivery as early-onset (<34 weeks), preterm (<37 weeks), or term (≥37 weeks).

SECONDARY OUTCOMES:
Sensitivity, specificity, PPV and NPV | an average of up to 1 year
  This study aims to evaluate the predictive performance of the test for preterm preeclampsia (PE) and all PE, specifically assessing its sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Niu, Master, Principal Investigator — Shenzhen Maternity and Child Healthcare Hospital
Locations (6):
- China (6):
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen, Guangdong
  - the Eighth Affiliated Hospital, Shenzhen, Guangdong
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Women's Hospital, of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No